CLINICAL TRIAL: NCT03620500
Title: Balance and Vestibular Impairments in Children With Cochlear Implantation
Brief Title: Balance in Children With Cochlear Implants
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cathey Norton, Staff Physical Therapist, Vanderbilt University Medical Center
Other Study IDs: 171127
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-03

CONDITIONS: Cochlear Implants; Sensory-Neural Hearing Loss; Balance Disorder
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with Cochlear Implants: Children with sensory neural hearing loss who undergo cochlear implantation will be monitored to see if balance develops normally in this population
  Interventions: Behavioral: Gross motor and developmental balance testing

INTERVENTIONS:
Behavioral: Gross motor and developmental balance testing — Balance (Pediatric Balance Scale) and gross motor skill development (Peabody Developmental Motor Scales, 2nd edition). Quality of life will be assessed using the Life-H (Assessment of Life Habits).

SUMMARY:
Cochlear implantation is performed in children with sensorineural hearing loss to restore hearing. Fifty percent of children with sensory neural hearing loss, who are candidates for cochlear implant, have vestibular (inner ear) dysfunction prior to surgery. Anatomically, the cochlea, semicircular canals, and otolith organs are located in close proximity in the inner ear and any procedure in the cochlea may affect the vestibular system, resulting in subsequent balance impairment. In addition, the process of implantation often results in further suppression of vestibular function necessary to develop normal balance. Vestibular dysfunction predisposes these children to balance impairments that can affect the normal development of gross motor skills such as sitting, standing, and walking. These balance and gross motor deficits may predispose the child to difficulties with safe community participation resulting in lower quality of life for the child and family.

Evidence in the literature suggests that children with vestibular loss do not recover to the same levels as their peers, especially in the area of activities requiring vestibular input for balance.

The purpose of this descriptive study is to examine balance, vestibular function, and gross motor skills in children following cochlear implantation over a period of one year. Children, ages 1 year to 5 years will be tested post cochlear implant , and at 6 and 12 months subsequent to initial testing, using clinically based tests of vestibular impairment (head impulse test, post rotary nystagmus or head shake nystagmus), balance (Pediatric Balance Scale) and gross motor skill development (Peabody Developmental Motor Scales, 2nd edition). Quality of life will be assessed using the Life-H (Assessment of Life Habits).

ELIGIBILITY:
Inclusion Criteria:

1. The Child must be a child between 12 months and 71 months of age.
2. The child should have received a cochlear implant within the previous year.
3. The child should be able to stand unsupported for 4 seconds.
4. Follow simple one step directions.

Exclusion Criteria:

1. Uncontrolled seizures
2. Any physician-recommended activity limitations that would preclude performing activities in the testing protocol.
3. Testing will not occur when the child is or has been acutely ill (i.e. fever, ear infection, etc.) within the previous week.
4. The participant must not have a known medical or developmental diagnosis that impacts his or her motor skills (i.e.

cerebral palsy, Down Syndrome) -

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with sensory neural hearing loss who are candidates for cochlear implantation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2023-08-03 (Estimated); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Change in the Peabody Developmental Motor Scales | Baseline to 1 year
  The Peabody Development Motor Scale measures balance in children compared to peers. A percentile score compared to typically developing peers is measured. A percentile score based on developmental age from birth to 5 years, 11 months.

CONTACTS AND LOCATIONS:
Overall Officials: Cathey Norton, DPT, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided